CLINICAL TRIAL: NCT03218137
Title: Use of Adenosine to Determine the Electrophysiological Mechanism of Premature Ventricular Contractions
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1609017561
Record Dates: First submitted 2017-06-29; First posted 2017-07-14 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Premature Ventricular Contraction (PVC)
Keywords: Subjects; diagnosed
MeSH Terms: conditions — Ventricular Premature Complexes; Disease | interventions — Adenosine; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Adenosine/ Verapamil Arm (Other): Adenosine: 0.84 mg/kg IV (140 mcg/kg/minute IV for 6 minutes) Verapamil: 0.15 mg/kg IV
  Adenosine is known to terminate ventricular arrhythmias that are due to triggered activity (ref Lerman). To study the effects of adenosine on PVC, the investigators will administer Verapamil to slow down the heart initially and adenosine after catheters are introduced to patients who are being treated for symptomatic PVC and have consented to treatment with an invasive electrophysiology study and catheter ablation.
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — Adenosine: 0.84 mg/kg (140 mcg/kg/minute IV for 6 minutes) Verapamil 0.15 mg/kg
  Other Names: Verapamil 0.15 mg/kg

SUMMARY:
Unblinded, controlled, non-randomized, mechanistic study to determine whether physiological mechanisms underlying PVC are sensitive to adenosine. One hundred subjects undergoing clinically-indicated, standard-of-care cardiac electrophysiology study (EPS) procedure for PVCs will receive adenosine and/or verapamil to learn if their arrhythmias are inducible similarly to sustained ventricular tachycardia.

DETAILED DESCRIPTION:
The cellular mechanism of premature ventricular contractions (PVCs) is unknown. The investigators have previously observed that 5% of patients in the investigators electrophysiology laboratory with ventricular outflow tract PVCs have inducible sustained ventricular tachycardia (VT) that behaves in a manner similar to patients who present clinically with sustained ventricular tachycardia, i.e., sensitive to adenosine and triggered activity. This suggests that outflow arrhythmias may be a continuum of a single mechanism.

Adenosine is known to terminate ventricular arrhythmias that are due to triggered activity (ref Lerman). To study the effects of adenosine on PVC, the investigators will administer Verapamil to slow down the heart initially and adenosine after catheters are introduced to patients who are being treated for symptomatic PVC and have consented to treatment with an invasive electrophysiology study and catheter ablation. The investigators will observe if there is any effect of reduced PVC following adenosine administration.

The investigators hypothesize that PVC will be suppressed by exogenous adenosine and/or verapamil. The information from this study will elucidate the underlying cellular mechanism of this common arrhythmia. Such knowledge could potentially lead to developing therapeutic targets. Moreover, it will have potential clinical applications for inducing outflow tract PVCs/VT in patients whose arrhythmia is suppressed at the time of their invasive electrophysiology study.

Analysis of the Holter recording of premature ventricular contractions:

Analysis of the PVC coupling intervals can be helpful for delineating the mechanism of PVCs. Holter monitors are being obtained on these patients prior to ablation as part of standard of care. Holters monitors, if performed at our institution, will be analyzed in detail in a retrospective fashion. Holter reports from 1/1/2015 - 5/15/2019 will be reviewed.

Specifically, evaluating the time intervals between PVCs and normal heart beats may elucidate potential arrhythmia mechanism as triggered activity or modulated parasystole. Since a subject has approximately 100,000 heart beats in 24 hours, the Holter data have to be read by a converter file and outputted to an Excel file for our further analysis. The investigators do not have access to a converter file and it is not commercially available. The investigators will send the de-identified data to Dr. Mortara at UCSF. The investigators will then analyze the timing intervals among PVCs and normal heart beats. It should be noted that these Holters are obtained as part of a patient's normal evaluation and are not obtained for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of premature ventricular contractions (PVCs)
* Scheduled to undergo an electrophysiology study with the intention of performing cardiac ablation for the treatment of PVCs
* Male or female between the ages of 18 and 70 years
* Capable of giving informed consent

Exclusion Criteria:

* Any structural heart disease
* Coronary artery disease (≥ 70% stenosis)
* Current treatment with anti-arrhythmic drugs
* Pregnant
* Asthma (if administering adenosine)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effects of Adenosine on premature ventricular contractions (PVCs) as measured by EKG; | baseline
  The metrics that will be collected will be:
  * Baseline frequency of premature ventricular contractions (PVCs)
  * Frequency of premature ventricular contractions (PVCs) during adenosine administration
Effects of verapamil on premature ventricular contractions (PVCs) as measured by EKGs. | baseline
  The metrics that will be collected will be:
  * Baseline frequency of premature ventricular contractions (PVCs)
  * Frequency of premature ventricular contractions (PVCs) during verapamil administration

CONTACTS AND LOCATIONS:
Overall Officials: James E Ip, M.D, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No